CLINICAL TRIAL: NCT01074749
Title: OSAT: Optimal Sensing in Atrial Tachyarrhythmia's Study
Brief Title: Optimal Sensing in Atrial Tachyarrhythmia's Study
Acronym: OSAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis indicated that endpoints can not be analysed with current dataset.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-09-058-ND-LV
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Sick Sinus Syndrome; Paroxysmal Atrial Fibrillation
Keywords: AF; Automatic Mode Switch; FFRW; paroxysmal AF
MeSH Terms: conditions — Sick Sinus Syndrome; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optisense lead (Active Comparator): Patients with an Accent pacemaker and an OptiSense atrial lead
  Interventions: Device: Accent Pacemaker
- Tendril lead (Active Comparator): Patients with an Accent pacemaker and a Tendril atrial lead
  Interventions: Device: Accent Pacemaker

INTERVENTIONS:
Device: Accent Pacemaker — Implantation of pacemaker
  Other Names: Accent DR RF 2212 Pacemaker; OptiSense 1999 atrial lead

SUMMARY:
The aim of the study is the comparison of two different leads in their capabilities to detect episodes and duration of paroxysmal atrial fibrillation (AF) and atrial tachyarrhythmia (AT), and the rejection of far field sensing of the far field R-wave (FFRW).

DETAILED DESCRIPTION:
The aim of the study is the comparison of two different leads in their capabilities to detect episodes and duration of paroxysmal AF and AT and the rejection of far field sensing of the far field R-wave (FFRW). The study aims to evaluate the accuracy of the detection of atrial tachyarrhythmias (ATAs). An improved detection can potentially increase the accuracy of clinical treatment decisions, based on device derived data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with class I or II pacing indications for Sick Sinus Syndrome with suspected paroxysmal atrial tachyarrhythmias over the last 6 months
* Signed informed consent
* Age >18 yrs

Exclusion Criteria:

* Severe valvular heart disease (echocardiogram less than 6 months old)
* Angina Pectoris class ≥ III
* Congestive heart failure - NYHA class ≥ III
* Left Ventricular Ejection Fraction < 35% (less than 6 months old)
* Hypertrophic Cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2010-07; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of undersensing of paroxysmal AF and AT from Holter recording. | 1-3 months

SECONDARY OUTCOMES:
Number and duration of inappropriate mode switches due to FFRW sensing during sinus rhythm. | 1-3 months

CONTACTS AND LOCATIONS:
Overall Officials: Willem De Voogt, MD PhD, Principal Investigator — St Lucas Andreas Hospital Amsterdam, Netherlands
Locations (1):
- Lucas Andreas Ziekenhuis, Amsterdam, Netherlands

REFERENCES:
- [Derived] Pakarinen S, Lehto M, Ruiter J, de Voogt WG. Enhanced detection of atrial tachyarrhythmias with pacing devices by using more accurate atrial sensing. J Interv Card Electrophysiol. 2022 Apr;63(3):601-609. doi: 10.1007/s10840-021-01066-z. Epub 2021 Oct 1. PMID 34599455